CLINICAL TRIAL: NCT00002523
Title: FOUR ARMS PHASE III CLINICAL TRIAL FOR T3-T4 RESECTABLE RECTAL CANCER COMPARING PRE-OPERATIVE PELVIC IRRADIATION TO PRE-OPERATIVE IRRADIATION COMBINED WITH FLUOROURACIL AND LEUCOVORIN WITH OR WITHOUT POST-OPERATIVE ADJUVANT CHEMOTHERAPY
Brief Title: Radiation Therapy, Surgery, and Chemotherapy in Treating Patients With Rectal Cancer That Can Be Surgically Removed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-22921; EORTC-22921
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug, giving the drugs in different ways, and combining radiation therapy and surgery with chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare radiation therapy alone before surgery with radiation therapy plus fluorouracil and leucovorin before surgery, with and without fluorouracil and leucovorin after surgery in patients with rectal cancer that can be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free and overall survival in patients with resectable adenocarcinoma of the rectum treated with preoperative radiotherapy with or without preoperative fluorouracil (5-FU) combined with leucovorin calcium (CF) and/or postoperative 5-FU/CF.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, sex, tumor location (0-5 vs 6-10 vs 11-15 cm from anal margin), and stage (T3 vs T4). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients undergo involved-field radiotherapy 5 days a week for 5 weeks followed 3-10 weeks later by abdominoperineal resection or anal-sparing resection according to local practice in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo radiotherapy as in arm I beginning on day 1 and leucovorin calcium (CF) IV followed by fluorouracil (5-FU) IV (1 hour before radiotherapy) on days 1-5 and 29-33, followed 3-10 weeks later by resection as in arm I in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients undergo radiotherapy followed 3-10 weeks later by resection as in arm I. Within 3-10 weeks after resection, patients receive CF followed by 5-FU on days 1-5. Chemotherapy continues every 4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm IV: Patients undergo preoperative radiotherapy with concurrent chemotherapy followed by resection as in arm II and postoperative chemotherapy as in arm III.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 992 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed resectable adenocarcinoma of the rectum

  * Any grade
  * Tumor macroscopically within 15 cm of anal margin on rigid rectoscopy
  * Tumor tethered or partially fixed on digital rectal exam and/or T3-4 on rectal ultrasound
* No acute or subacute bowel obstruction without colostomy diversion
* No chronic inflammatory disease of the ileum and/or colon
* No primary adenocarcinoma of the anal canal
* No distant metastasis

PATIENT CHARACTERISTICS:

Age:

* 80 and under

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count greater than 2,000/mm^3
* Platelet count greater than 130,000/mm^3

Hepatic:

* Not specified

Renal:

* Creatinine less than 1.36 mg/dL

Cardiovascular:

* No angina pectoris

Other:

* No other prior malignancy except basal cell skin cancer or carcinoma in situ of the uterine cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for adenocarcinoma of the rectum

Chemotherapy

* No prior chemotherapy for adenocarcinoma of the rectum

Endocrine therapy

* No prior endocrine therapy for adenocarcinoma of the rectum

Radiotherapy

* No prior radiotherapy for adenocarcinoma of the rectum

Surgery

* No prior surgery for adenocarcinoma of the rectum

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1011 (Actual)
Dates: Start 1993-04; Primary Completion 2003-03 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Bosset, MD, Study Chair — Hopital Jean Minjoz
Locations (35):
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Hopital Civil de Charleroi, Charleroi
  - Centre Hospitalier Universitaire de Tivoli, La Louvière
  - Clinique Sainte Elisabeth, Namur
- France (18):
  - Centre Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier General, Belfort
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - C.H.U. de Brest, Brest
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - CHR de Grenoble - La Tronche, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Service Cancerologie Polyclinique Clairval, Marseille
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Clinique De Valdegour, Nîmes
  - Hopital Jean Bernard, Poitiers
  - Clinique Sainte Clotilde, Sainte Clotilde
  - Centre Paul Strauss, Strasbourg
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Saint-Yves, Vannes
- Krankenhaus des Kreises Hameln-Pyrmont, Hamelin, Germany
- Rambam Medical Center, Haifa, Israel
- Netherlands (2):
  - University Medical Center Nijmegen, Nijmegen
  - Dr. Bernard Verbeeten Instituut, Tilburg
- Medical University of Gdansk, Gdansk, Poland
- Institute of Oncology and Radiology of Serbia, Belgrade, Serbia
- Spain (3):
  - Hospital General Universitari Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia - Hospital Duran i Reynals, Barcelona
  - Hospital General Gregorio Maranon, Madrid
- Switzerland (2):
  - Kantonsspital Basel, Basel
  - UniversitaetsSpital, Zurich
- Dokuz Eylul University School of Medicine, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Bonnetain F, Bosset J, Gerard J, et al.: An analysis of preoperative chemoradiotherapy with 5FU/leucovorin for T3-4 rectal cancer on survival in a pooled analysis of EORTC 22921 and FFCD 9203 trials: surrogacy in question? [Abstract] J Clin Oncol 29 (Suppl 15): A-3506, 2011.
- [Background] den Dulk M, Putter H, Collette L, Marijnen CAM, Folkesson J, Bosset JF, Rodel C, Bujko K, Pahlman L, van de Velde CJH. The abdominoperineal resection itself is associated with an adverse outcome: the European experience based on a pooled analysis of five European randomised clinical trials on rectal cancer. Eur J Cancer. 2009 May;45(7):1175-1183. doi: 10.1016/j.ejca.2008.11.039. Epub 2009 Jan 6. PMID 19128956
- [Result] Monnien F, Zaki H, Borg C, Mougin C, Bosset JF, Mercier M, Arbez-Gindre F, Kantelip B. Prognostic value of phosphorylated STAT3 in advanced rectal cancer: a study from 104 French patients included in the EORTC 22921 trial. J Clin Pathol. 2010 Oct;63(10):873-8. doi: 10.1136/jcp.2010.076414. PMID 20876317
- [Result] Tiv M, Puyraveau M, Mineur L, Calais G, Maingon P, Bardet E, Mercier M, Bosset JF. Long-term quality of life in patients with rectal cancer treated with preoperative (chemo)-radiotherapy within a randomized trial. Cancer Radiother. 2010 Oct;14(6-7):530-4. doi: 10.1016/j.canrad.2010.06.017. Epub 2010 Aug 24. PMID 20797891
- [Result] Collette L, Bosset JF, den Dulk M, Nguyen F, Mineur L, Maingon P, Radosevic-Jelic L, Pierart M, Calais G; European Organisation for Research and Treatment of Cancer Radiation Oncology Group. Patients with curative resection of cT3-4 rectal cancer after preoperative radiotherapy or radiochemotherapy: does anybody benefit from adjuvant fluorouracil-based chemotherapy? A trial of the European Organisation for Research and Treatment of Cancer Radiation Oncology Group. J Clin Oncol. 2007 Oct 1;25(28):4379-86. doi: 10.1200/JCO.2007.11.9685. PMID 17906203
- [Result] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Result] Bosset J, Calais G, Mineur L, et al.: Preoperative radiotherapy in rectal cancer: role and place of fluorouracil-based chemotherapy. Final results of the EORTC 22921 phase III trial. [Abstract] American Society of Clinical Oncology 2005 Gastrointestinal Cancers Symposium, 27-29 January 2005, Miami, Florida. A-255, 2005.
- [Result] Bosset JF, Calais G, Mineur L, et al.: Preoperative radiation (Preop RT) in rectal cancer: effect and timing of additional chemotherapy (CT) 5-year results of the EORTC 22921 trial. [Abstract] J Clin Oncol 23 (Suppl 16): A-3505, 247s, 2005.
- [Result] Bosset JF, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Briffaux A, Collette L. Enhanced tumorocidal effect of chemotherapy with preoperative radiotherapy for rectal cancer: preliminary results--EORTC 22921. J Clin Oncol. 2005 Aug 20;23(24):5620-7. doi: 10.1200/JCO.2005.02.113. Epub 2005 Jul 11. PMID 16009958
- [Result] Bosset JF, Calais G, Mineur L, et al.: Does the addition of chemotherapy (CT) to preoperative radiotherapy (preopRT) increase the pathological response in patients with resected rectal cancer: report of the 22921 EORTC phase III trial. [Abstract] J Clin Oncol 22 (Suppl 14): A-3504, 246, 2004.
- [Result] Bosset JF, Calais G, Daban A, et al.: Does the addition of chemotherapy to preoperative radiation increase acute toxicity in patients with rectal cancer: report of 22921 EORTC phase III trial . [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1179, 2003.
- [Result] Kouloulias VE, Bosset JF, van Tienhoven G, Davis BJ, Pierart M, Poortmans P; EORTC Radiotherapy Group. European Organization for Research and Treatment of Cancer. Quality assurance in the EORTC 22921 trial on preoperative radiotherapy with or without chemotherapy for resectable rectal cancer: evaluation of the individual case review procedure. Eur J Cancer. 2002 Sep;38(14):1849-56. doi: 10.1016/s0959-8049(02)00174-0. PMID 12204666
- [Derived] Bosset JF, Calais G, Mineur L, Maingon P, Stojanovic-Rundic S, Bensadoun RJ, Bardet E, Beny A, Ollier JC, Bolla M, Marchal D, Van Laethem JL, Klein V, Giralt J, Clavere P, Glanzmann C, Cellier P, Collette L; EORTC Radiation Oncology Group. Fluorouracil-based adjuvant chemotherapy after preoperative chemoradiotherapy in rectal cancer: long-term results of the EORTC 22921 randomised study. Lancet Oncol. 2014 Feb;15(2):184-90. doi: 10.1016/S1470-2045(13)70599-0. Epub 2014 Jan 17. PMID 24440473